CLINICAL TRIAL: NCT00289172
Title: A Multicenter Study of the Immunogenicity & Safety of 2 Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus Vaccine (RIX4414) as Primary Dosing of Healthy Infants in India Aged Approximately 8 Wks at the Time of the First Dose
Brief Title: Assess the Immunogenicity & Safety of 2 Doses of Oral Live Attenuated Human Rota(HRV)Vaccine in Healthy Infants in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 103792
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections

INTERVENTIONS:
Biological: Live attenuated human rotavirus vaccine

SUMMARY:
Rotavirus disease is the most common cause of gastroenteritis and dehydration in young children worldwide. The global public health burden has prompted the development of a human rotavirus vaccine against rotavirus disease by GlaxoSmithKline Biologicals. This pre-registration study is undertaken to provide immunogenicity, reactogenicity and safety data for the vaccine when used in Indian infants aged approximately 8 weeks at the time of the first dose.

DETAILED DESCRIPTION:
The study consists of two groups of children to be recruited in different centers in India. One group will receive the HRV vaccine and one group will receive the placebo. The vaccine or placebo will be administered starting at 8-12 weeks of age, according to a two dose schedule (0, 1 months schedule). The study will consist of three visits. A 8-day (Day 0 - 7) follow-up period will be observed for general symptoms solicited in the study. A 31-day (Day 0 - 30) follow-up will be observed for other unsolicited symptoms. Serious adverse events (SAEs) will be followed-up throughout the study. A stool sample will be collected from the child at any point during the study if he/ she develops any GE.

ELIGIBILITY:
"Inclusion criteria:

* A male or female between, and including, 8 and 10 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* The subjects should have been administered the first dose of DTP/ OPV/ hepatitis B vaccines as per the local universal immunization program at 6 weeks of age.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine or the routine UIP vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth. (For corticosteroids, this will mean prednisone, or equivalent, >= 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Any chronic drug therapy to be continued during the study period.
* Administration of a vaccine not foreseen by the study protocol within 6 weeks of the first dose of vaccine or planned administration during the study of a vaccine not foreseen by the study protocol, with the exception of diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b (Hib), OPV and vaccination against tuberculosis, which can be given with at least two weeks separation from the first and subsequent dose of the study vaccine.
* Prior administration of experimental rotavirus vaccine.
* History of confirmed rotavirus gastroenteritis.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the GI tract or other serious medical condition as determined by the investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection based on physical examination (no laboratory testing is required).
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Gastroenteritis (diarrhea) within 7 days preceding the study vaccine administration (warrants deferral of the vaccination).
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or medical history.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period. Oral intake of immunoglobulins via breastfeeding is allowed.

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360
Dates: Start 2006-02-10; Study Completion 2006-09-08 (Actual)

PRIMARY OUTCOMES:
Percentage of seroconversion (anti-rota serum IgA) in children, after two doses of HRV vaccine versus two doses of placebo.

SECONDARY OUTCOMES:
Fever, vomiting, diarrhea. Solicited symptoms. Unsolicited events. SAEs. Presence of rotavirus in GE stools.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- India (4):
  - GSK Investigational Site, Chandigarth
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Vellore

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bhattacharya SK et al. Immune response in infants sero-positive at pre-vaccination human rotavirus vaccine Rotarix™. Poster presented at WSPID, Bangkok, Thailand,15-18 November 2007
- [Background] Bose et al. Safety and immunogenicity of RIX4414 (Rotarix TM) live-attenuated human rotavirus vaccine in Indian infants. Poster presented at WSPID, Bangkok, Thailand, 15-18 November 2007.
- [Background] Narang A, Bose A, Pandit AN, Dutta P, Kang G, Bhattacharya SK, Datta SK, Suryakiran PV, Delem A, Han HH, Bock HL. Immunogenicity, reactogenicity and safety of human rotavirus vaccine (RIX4414) in Indian infants. Hum Vaccin. 2009 Jun;5(6):414-9. doi: 10.4161/hv.5.6.8176. Epub 2009 Jun 15. PMID 19276664
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 103792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103792 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register